CLINICAL TRIAL: NCT01000610
Title: An Open Label Study to Evaluate the Safety and Efficacy of Rituximab in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Prior Treatment With Methotrexate
Brief Title: A Study of MabThera (Rituximab) in Patients With Rheumatoid Arthritis and an Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20549
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate; Methylprednisolone

ARMS (1):
- single arm (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: methotrexate; Drug: methylprednisolone

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1000 mg iv infusion on days 1 and 15
Drug: methotrexate — 10-25 mg weekly (oral or parenteral)
Drug: methylprednisolone — 100 mg iv prior to each rituximab infusion

SUMMARY:
In this open-label single arm study the safety and efficacy of Mabthera will be evaluated in patients with active rheumatoid arthritis who have had an inadequate response to methotrexate. Patients will receive MabThera (1000mg iv infusion) on days 1 and 15, and background methotrexate (10-25mg po or sc weekly). After the initial study period of 24 weeks, eligible patients may receive up to 3 re-treatments with MabThera. The anticipated time on study treatment is 1-2 years and target sample size is <50

ELIGIBILITY:
Inclusion Criteria:

* adult patients >/= 18 years of age
* rheumatoid arthritis DAS28 >/= 3.2
* receiving treatment on an outpatient basis
* experienced an inadequate response to previous or current treatment with methotrexate

Exclusion Criteria:

* rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA
* history of or current inflammatory joint disease other than RA
* previous treatment with any cell-depleting therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-03-17 (Actual); Primary Completion 2012-05-16 (Actual); Study Completion 2012-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Tunisia (4):
  - Hopital Farhat Hached; Service Rhumatologie, Sousse
  - Hopital Charles Nicole; Service Rhumatologie, Tunis
  - Hopital La Rabta; Service Rhumatologie, Tunis
  - Hopital Mongi Slim; Service Rhumatologie, Tunis

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Participants received rituximab 1000 milligrams (mg) intravenous (iv) infusion on Days 1 and 15 along with methotrexate 10-25 mg weekly, orally or parenterally. Participants could receive concomitant treatment with corticosteroids (less than or equal to [≤] 10 milligrams per day (mg/day) prednisone or equivalent) or intra-articular corticosteroids, non-steroid anti-inflammatory drugs (NSAIDs) and analgesics throughout the study period at the discretion of the investigator. All participants received methylprednisolone100 mg iv prior to each rituximab infusion.
Period: Overall Study
Arm/Group | Rituximab
Started | 18
Completed | 12
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 4
Not completed — Treatment failure | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population: All participants who received any part of an infusion have been included in the ITT analysis. Participants who prematurely withdrew from the study for any reason and for whom an assessment was not performed for whatever reason, were still included in the ITT analyses.
Groups:
- Rituximab: Participants received rituximab 1000 mg iv infusion on Days 1 and 15 along with methotrexate 10-25 mg weekly, orally or parenterally. Participants could receive concomitant treatment with corticosteroids (≤ 10 mg/day prednisone or equivalent) or intra-articular corticosteroids, NSAIDs and analgesics throughout the study period at the discretion of the investigator. All participants received methylprednisolone 100 mg iv prior to each rituximab infusion.
Arm/Group | Rituximab
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events (AEs)
Time Frame: Days 1 and 15, every 8 weeks up to Week 24 and and then every 3 months up to 18 months for a total of 104 weeks
Population: Safety Population: Included all participants who have received any part of an infusion of study medication.
Measure: Number; unit: number of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 18
number of participants
  Participants who experienced an AE | 11
  Participants who experienced more than 1 AE | 7

2. Secondary Outcome: Percentage Change in Disease Activity Score 28 (DAS28) From Baseline to Week 24
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], participant's global assessment of disease activity [visual analog scale: [VAS] 0 equals (=) no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to 10. Scores less than (<) 2.6 indicate best disease control and scores greater than or equal to (≥) 5.1 indicate worse disease control. DAS28 Remission is defined as a DAS28 score < 2.6. The average improvement at each visit to the group score is equal to the formula (Previous DAS28 minus [-] current DAS 28)/ Previous DAS 28 x 100. Negative percentages indicate that the participant has worsened in comparison to last evaluation, and positive percentages indicate improvement of its DAS28 score and correlated with a bettering of clinical situation.
Time Frame: Baseline and Week 24
Population: ITT population; Only participants with DAS28 values at both Baseline and Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Rituximab
Number analyzed (Participants) | 16
percentage change from baseline | -1.7 (49.4)

3. Secondary Outcome: Percentage of Participants Whose DAS28 Improved by >1.2 at Week 24
Description: The DAS28 score is a measure of the participant's disease activity calculated using the TJC [28 joints], SJC [28 joints], participant's global assessment of disease activity [VAS: 0 = no disease activity to 100 = maximum disease activity] and the ESR for a total possible score of 0 to 10. Scores < 2.6 indicate best disease control and scores ≥ 5.1 indicate worse disease control. DAS28 Remission is defined as a DAS28 score < 2.6. An improvement of >1.2 was considered to be clinically significant improvement.
Time Frame: Baseline and Week 24
Population: ITT population; Only participants with DAS28 values at both Baseline and Week 24 were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 16
percentage of participants | 75.0

4. Secondary Outcome: Change in Bone Density (in Participants Untreated With Bisphosphonates)
Description: Bone mineral density test was performed using x-ray radiation and the values of bone density were provided directly by the apparatus as grams per square centimeter (g/cm^2) . T-score is the number of standard deviations above or below the mean for a healthy 30 year old adult of the same sex and ethnicity as the participant. A T-score with above -1 is normal bone density level. A T-score between -1 and -2.5 means that the bone density is below normal and it might be a sign of an osteopenia and may also lead into osteoporosis. A T-score below -2.5 indicates osteoporosis.
Time Frame: Screening and Week 84
Population: ITT population; only participants with an assessment at both screening and Week 84 were included in the analysis.
Measure: Number; unit: t-score
Arm/Group | Rituximab
Number analyzed (Participants) | 1
t-score
  Screening | -1.82
  Week 84 | -1.6

ADVERSE EVENTS:
Time Frame: AEs were recorded from the day of first infusion until the End of Study at 104 weeks.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 6/18
Other Adverse Events (participants affected / at risk) | 9/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=18)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Persistent thrombopenia (Blood and lymphatic system disorders) | 1
Rectal bleeding (Gastrointestinal disorders) | 1
Ventricular Extra systolebigeminy (Cardiac disorders) | 1
Severe infusion reaction (Injury, poisoning and procedural complications) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=18)
Blurred Vision (Eye disorders) | 1
Hyperglycemia (Endocrine disorders) | 1
Multi-sensitive Streptococcus Cystitis (Infections and infestations) | 1
Hypertension (Blood and lymphatic system disorders) | 2
Keratitis Secca (Skin and subcutaneous tissue disorders) | 1
Red Throat (General disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Somnolence (General disorders) | 1
Influenza (Infections and infestations) | 1
Muscular Pain (Musculoskeletal and connective tissue disorders) | 1
Nocturnal Sweating (General disorders) | 1
Headache (General disorders) | 1
Dyspnea Stage 2 (Respiratory, thoracic and mediastinal disorders) | 1
Productive Cough-Yellow Expectorations (Respiratory, thoracic and mediastinal disorders) | 1
Pneumopathy Infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.